CLINICAL TRIAL: NCT01005875
Title: RAD 0901- Stereotactic Radiation Therapy and Sorafenib in the Treatment of Hepatocellular Carcinoma
Brief Title: Stereotactic Radiation Therapy and Sorafenib in the Treatment of Hepatocellular Carcinoma
Acronym: RAD 0901
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor(Bayer)did not wish to continue with study due to slow accrual. Therefore, there is insufficient data and will not be any study results/outcomes.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Kimberly Keene, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F090910004
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Hepatocellular carcinoma; HCC; Liver Cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation followed by Sorafenib (Experimental): Radiation therapy, stereotactic body radiation therapy followed by Sorafenib
  Interventions: Drug: Sorafenib; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Sorafenib — Nexavar in bottles of 120 tables
  Other Names: BAY 43-9006; Nexavar
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT

SUMMARY:
This study is to determine the safety and efficacy of stereotactic body radiotherapy (SBRT) and treatment drug in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A or B7 cirrhosis.
* No prior radiation therapy to the upper right abdominal quadrant.
* Size of each tumor less than 6 cm.
* Three or less known lesions.
* More than 800 cc of uninvolved liver.
* Age > 19 years old
* ECOG Performance Status 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following:
* Hemoglobin > 8.5 g/dl
* Platelet count > 50,000/mm3
* Total bilirubin < 1.5 times ULN
* ALT and AST < 2.5 times the ULN ( < 5 x ULN for patients with liver involvement)
* Creatinine < 1.5 times ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Child-Pugh class B8 or C cirrhosis.
* ECOG greater than or equal to 2.
* Uncontrolled ascites despite medical management.
* Less than 800 cc of uninvolved liver.
* Prior radiotherapy to the upper abdominal quadrant.
* Prior antiangiogenic or tyrosine kinase inhibitor therapy Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina(anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure >90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Pregnant or lactating female.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S Keene, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Followed by Sorafenib
Started | 5
Completed | 2
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 60 [50 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Determine the Safety and Tolerability of Sequential SBRT and Sorafenib in Patients With Unresectable Hepatocellular Carcinoma
Description: Number of subjects experiencing a Grade 5 toxicity related to SBRT and sorafenib
Time Frame: between baseline and 3 years
Measure: Number; unit: participants
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: The Degree of Change in Necrosis and Vascular Permeability Via Dynamic Contrast Enhanced (DCE) and Diffusion-weighted Imaging (DWI) Magnetic Resonance Imaging (MRI) as Measured by Tumor Volume
Description: mean tumor volume at baseline, 4 weeks and 10 weeks after start of treatment
Time Frame: baseline, 4 weeks and 10 weeks
Measure: Mean (Standard Deviation); unit: centimeters^3
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 2
centimeters^3
  at baseline | 98 (71)
  at 4 weeks after baseline | 65 (42)
  at 10 weeks after baseline | 22 (8)

3. Secondary Outcome: The Degree of Change in Necrosis and Vascular Permeability Via Dynamic Contrast Enhanced (DCE) and Diffusion-weighted Imaging (DWI) Magnetic Resonance Imaging (MRI) as Measured by Ktrans (Volume Transfer Coefficient).
Description: The initial mean Ktrans at baseline, 4 weeks and 10 week. K trans is used to describe the uptake of gadolinium contrast in tissue.
Time Frame: baseline, 4 weeks and 10 weeks
Measure: Mean (Standard Deviation); unit: min^ -1
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 2
min^ -1
  at baseline | 0.022 (0.009)
  at 4 weeks after baseline | 0.017 (0.009)
  at 10 weeks after baseline | 0.014 (0.006)

4. Secondary Outcome: The Degree of Change in Necrosis and Vascular Permeability Via Dynamic Contrast Enhanced (DCE) and Diffusion-weighted Imaging (DWI) Magnetic Resonance Imaging (MRI) as Measured by Kep. Kep Describes How Fast Contrast Can Redistribute in Tissue.
Description: The Kep as measures by MRI at baseline, 4 weeks after baseline, and 10 weeks after baseline.
Time Frame: baseline, 4 weeks after baseline and 10 weeks post baseline
Measure: Mean (Standard Deviation); unit: Min^ -1
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 2
Min^ -1
  at baseline | 0.062 (0.018)
  at 4 weeks after baseline | 0.053 (0.013)
  at 10 weeks after baseline | 0.050 (0.014)

5. Secondary Outcome: The Degree of Change in Necrosis and Vascular Permeability Via Dynamic Contrast Enhanced (DCE) and Diffusion-weighted Imaging (DWI) Magnetic Resonance Imaging (MRI) as Measured by ADC (Apparent Diffusion Coefficient).
Description: the measured ADC at baseline, 4 weeks after baseline and then 10 weeks after baseline. ADC quantifies the motion of water protons from an MRI.
Time Frame: baseline, 4 weeks post baseline, 10 weeks post baseline
Measure: Mean (Standard Deviation); unit: milimeters^2/sec
Arm/Group | Radiation Followed by Sorafenib
Number analyzed (Participants) | 2
milimeters^2/sec
  at baseline | 1.29 (0.09)
  at 4 weeks after baseline | 1.55 (0.13)
  at 10 weeks after baseline | 1.65 (0.18)

ADVERSE EVENTS:
Time Frame: Baseline and 3 years
Arm/Group | Radiation Followed by Sorafenib
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Followed by Sorafenib (N=5)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Followed by Sorafenib (N=5)
Nausea (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed due to slow accural and enrolled 5 of the 10 planned patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes